CLINICAL TRIAL: NCT06026722
Title: "Behavioral and Cognitive Therapy for Insomnia in the Treatment of Pathological Gambling: Randomised and Control Pilot Study
Brief Title: Behavioral and Cognitive Therapy for Insomnia in the Treatment of Pathological Gambling
Acronym: SOMJEU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP221164; 2023-A00397-38 (Other: IDRCB)
Record Dates: First submitted 2023-06-14; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-06

CONDITIONS: Gambling Disorder Treatment
Keywords: Gambling disorder,sleep disorder, insomnia, CBT-I, addiction
MeSH Terms: conditions — Gambling; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Behavior, Addictive | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): patient will follow cognitive behavioral therapy for insomnia 1 per week during 1 month. this therapy will start a month after inclusion.
  Interventions: Behavioral: cognitive behavioral therapy for insomnia
- control group (waiting list) (Other): patient will follow cognitive behavioral therapy for insomnia 1 per week during 1 month. this therapy will start 7 month after inclusion.
  Interventions: Behavioral: cognitive behavioral therapy for insomnia

INTERVENTIONS:
Behavioral: cognitive behavioral therapy for insomnia — CBT-I is a 4-session program built around 3 main axes: psychoeducation on sleep hygiene, cognitive therapy and behavioral stimulus control, sleep restriction and relaxation. Each of the 3 axes will be worked on over 3 sessions, the last one being a summary and consolidation session of the first 3. For ethical reasons, it has been decided that patients in the control arm will also follow CBT-I (on a waiting list). The control group will have the same follow-up as the experimental group, but will start the intervention 6 months after the experimental group. This will enable all patients to access CBT-I.

SUMMARY:
Gambling is a public health risk. The wide panel of games available (poker, sport bets, scratch card games, slot machines, stock speculation …) and the advent of the Internet means that this behaviour is increasingly monitored on an epidemiological level, to the point where its pathological practice is now recognized in the DSM-5. Indeed, the scientific literature suggests a bidirectional link between use disorders and sleep disorders.

Sleep deprivation is known to lead to impaired judgment (risk-taking), increased sensitivity to reward, attentional difficulties and poor emotional management. The reverse has also been demonstrated: for example, playing at night has an impact on sleep quality, particularly in terms of difficulty falling asleep, ruminations about the game and a delay in the sleep-wake phase. Sleep disorders also affect patients undergoing withdrawal and/or cessation of a substance or behavior. This established link between addictions and circadian rhythms is important, since it is suggested that patients who are more impaired in both respects are more likely to relapse and respond less well to treatment.

In addictology, Behavioral and Cognitive Therapy for Insomnia (CBT-I) has proved effective in alcohol-dependent subjects in four studies. All reported a better quality of life (less depressive cognitions, better lifestyle) after CBT-I, although only one study reported a numerical reduction in consumption.The treatment of substance use disorders (AUD) remains limited : no pharmacological treatment has proved its worth, and the reference treatment remains mainly CBT. Despite the indisputable effectiveness of CBT, between 14% and 50% of patients are reported to have broken off from follow-up and care, and almost 90% of patients end up relapsing.

DETAILED DESCRIPTION:
Gambling is a public health risk. The wide panel of games available (poker, sports betting, scratch cards, slot machines, even stock market speculation...) and the advent of the Internet mean that this behavior is increasingly monitored from an epidemiological point of view, to the extent that its pathological practice is now recognized in the DSM-5. The DSM-5 characterizes the disorder as maladaptive (i.e., a loss of control leading to negative consequences for daily life), persistent (i.e., to the point of obsessive thoughts about it, and returning to it to "chase losses") and repeated (i.e., the need to play more and more to feel the initial effects) gambling. The Internet has made it possible to access gambling day and night, in complete anonymity, removing any inhibitions and facilitating dematerialized gambling, which is less palpable but just as damaging for patients. According to the "Observatoire des Jeux en France" in 2019, 6% of the French population could be problem gamblers (4.4% at moderate risk, and 1.6% pathological gamblers). Although prohibited for minors, gambling is becoming increasingly democratized among younger populations, and among 17-year-olds who gambled at least once in the year of 2017, 1.6% could be pathological gamblers. According to the e-Games France 2017 survey, being male (OR=1.57), young (OR=6.64), rather educated (OR=2.83), not retired (active, unemployed or student) (OR=26.8), with low income (OR=2.86) are socio-demographic characteristics linked to a higher risk of problem gambling. Moreover, according to the same survey, Internet gambling is more risky than "traditional" gambling, with 9.4% of online gamblers presenting a problem (compared with 0.9% of traditional gamblers) and 13% being pathological gamblers (compared with 3.9%). The health and social impact of online gambling in France remains poorly described, due to the marginalization of gambling disorders (few specialists, "shameful" addiction) and limited access to care. The impact on individuals and their families can be considerable, with financial consequences at the top of the list, including over-indebtedness and bankruptcy. The difficulties can also be relational and familial (separations, isolation, etc.), professional (redundancy, loss of opportunity, etc.), psychological (depression, anxiety, suicide, etc.) or physical (asthenia, symptoms linked to the consumption of alcohol or other psychoactive products, etc.). Scientific literature also suggests a so-called bidirectional link between use disorders and sleep disorders. Sleep deprivation is known to lead to impaired judgment (risk-taking), heightened sensitivity to reward, attentional difficulties and poor emotional management.

The reverse has also been demonstrated: for example, playing at night has an impact on sleep quality, particularly in terms of difficulty falling asleep, ruminations about the game and a delay in the sleep-wake phase. Sleep disorders also affect patients undergoing withdrawal and/or cessation of a substance or behavior. This established link between addictions and circadian rhythms is important, since it is suggested that patients who are more impaired in both respects are more likely to relapse and respond less well to treatment.

Three studies looked briefly at the perceived subjective sleep quality of pathological gamblers (by asking them whether they slept well, yes or no) and also observed more degraded sleep in gamblers compared to controls. Another study found a positive correlation between pathological gambling severity, difficulty falling asleep and poor sleep hygiene.

A larger U.S.-based study (N=3435) also reported that pathological gamblers were significantly more likely to report one or all of three insomnia criteria (difficulty falling asleep, daytime sleepiness, and early waking). Two more recent studies also point in this direction: an Australian study found an association between the DSM-5 diagnosis of insomnia, sleep of poor quality judged by the patient, and the severity of pathological gambling. According to a Canadian study of online poker players, the most sleep-deprived players were the most exposed to financial losses and a greater number of hands played in equal playing time. Other studies even suggest an indirect link between sleep and pathological gambling during periods of extreme stress. The stress of continual losses is associated with poor sleep quality, and between-games phases (i.e., withdrawal) are subject to intense stress, with negative effects on sleep. Finally, on a more objective level, actimetry data revealed poor sleep quality (shortened nights, "non-restorative" sleep, longer sleep times, multiple awakenings) in addicted patients. Given the addictive potential of most hypnotic pharmacological treatments, treating sleep disorders in an addicted patient is always a delicate matter.

However, no study has investigated the therapeutic effect of non-pharmacological treatment of sleep disorders in pathological gamblers.

Behavioral and Cognitive Therapy for Insomnia (CBT-I) is considered the gold standard for the treatment of sleep disorders. CBT-I has 3 main components: psycho-education on sleep hygiene, cognitive therapy and behavioral therapy on stimulus control, sleep restriction and relaxation.

This non-pharmacological intervention has proved effective in improving sleep, fatigue and quality of life in subjects suffering from chronic insomnia, up to 3 years after CBT-I (insomnia severity score ISI down from 18.6 to 13 after CBT-I, with improvement to 11.9 p<0.001 after 3 years in 90% of patients).

In addictology, this therapy has proved effective in alcohol-dependent subjects in four studies. All reported a better quality of life (less depressive cognitions, better lifestyle) after CBT-I, although only one study reported a numerical reduction in consumption.The treatment of substance use disorders (AUD) remains limited : no pharmacological treatment has proved its worth, and the reference treatment remains mainly CBT. Despite the indisputable effectiveness of CBT, between 14% and 50% of patients are reported to have broken off from follow-up and care, and almost 90% of patients end up relapsing.

ELIGIBILITY:
Inclusion Criteria:

* Patient with criteria of chronic gambling disorder according to DSM-5 defined as score greater than or equal to 5 for th South Oaks Gamling Screen (SOGS) and insomnia according to DSM-5 with score at ISI greater than 10.
* Outpatient or day hospitalization for gambling disorder in one of the psychiatric departments of the study centers for a period of care of at least 6 months.
* write, read and speak French
* Affiliated to a social security scheme (excluding State Medical Aid)
* volonteer, able to give their consent, informed

Exclusion Criteria:

* Specially protected adult, under guardianship or curatorship, or under therapeutic injunction
* pregnant woman
* Presence of any psychiatric pathology or clinically significant or unstable psychiatric appearance (decompensated bipolar disorder, decompensated schizophrenia, neurodegenerative disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
variation of the severity of gambling disorder betwen day 0 and month 4 of inclusion | day 0, month 4 of inclusion
  difference of G-SAS (gambling symptom assessment scale) score between day 0 and month 4

SECONDARY OUTCOMES:
variation of the severity of gambling disorder betwen day 0 and month 7 of inclusion | day 0, month 7 of inclusion
  difference of G-SAS score between day 0 and month 7
variation of the severity of gambling disorder during patient follow up | day0, month4, month 7 of inclusion
  difference of G-SAS score between day 0, month and month 7
variation of relative amplitude of rhythms betwen day 0 and month 7 of inclusion | day 0, month 7 of inclusion
variation of relative amplitude of rhythms betwen day 0 and month 4 of inclusion | day 0, month 4 of inclusion
variation of total sleep time betwen Day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
variation of total sleep time betwen Day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
variation wake after sleep onset (WASO) Day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
variation wake after sleep onset (WASO) betwen Day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
change of sleep fragmentation index betwen day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
change in sleep fragmentation index betwen day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
change in sleep efficiency index betwen day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
change in sleep efficiency index betwen day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
change of Insomnia Severity Index (ISI) score betwen day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
change of Insomnia Severity Index (ISI) score betwen day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
change of Pittsburg Sleep Quality Index (PSQI) score betwen day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
change of Pittsburg Sleep Quality Index (PSQI) score betwen day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
change of Munich Chronotype Type Questionnaire (MCTQ) score betwen day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
change of Munich Chronotype Type Questionnaire (MCTQ) score betwen day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
change of Epworth Sleepiness Scale (ESS) score betwen day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
change of Epworth Sleepiness Scale (ESS) score betwen day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
sleep fragmentation index betwen day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
sleep fragmentation index betwen day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
presume sleep time betwen day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
presume sleep time betwen day 0 and month 7 of inclusion | day 0 and month 7 of inclusion
time spend in bed betwen day 0 and month 4 of inclusion | day 0 and month 4 of inclusion
time spend in bed betwen day 0 and month 7 of inclusion | day 0 and month 7 of inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Bichat - Claude-Bernard hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No